CLINICAL TRIAL: NCT00872781
Title: An Open Label, Balanced, Randomized, Two-Treatment, Two-Period, Two-Sequence, Single-Dose, Crossover Bioavailability Study Comparing Fixed Dose Combination of Quinapril HCl 20 mg and Hydrochlorothiazide 25 mg Tablets of OHM Laboratories Inc (a Subsidiary of Ranbaxy Pharmaceuticals Inc) With ACCURETICTM Tablets (Containing Fixed Dose Combination of Quinapril HCl 20 mg and Hydrochlorothiazide 25 mg) of Parke Davis, in Healthy, Adult, Human, Male Subjects Under Fasting Condition.
Brief Title: Bioequivalence Study of Quinapril Hydrochloride 20 mg and Hydrochlorothiazide 25 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Laboratories
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 255_QUIHY_07
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Healthy
Keywords: Bioequivalence fixed dose combination of Quinapril HCl 20 mg and Hydrochlorothiazide 25 mg tablets
MeSH Terms: interventions — Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): fixed dose combination of Quinapril HCl 20 mg and Hydrochlorothiazide 25 mg tablets of OHM Laboratories Inc (a subsidiary of Ranbaxy pharmaceuticals Inc)
  Interventions: Drug: fixed dose combination of Quinapril HCl 20 mg and Hydrochlorothiazide 25 mg tablets
- 2 (Active Comparator): ACCURETICTM tablets (containing fixed dose combination of Quinapril HCl 20 mg and Hydrochlorothiazide 25 mg)
  Interventions: Drug: fixed dose combination of Quinapril HCl 20 mg and Hydrochlorothiazide 25 mg tablets

INTERVENTIONS:
Drug: fixed dose combination of Quinapril HCl 20 mg and Hydrochlorothiazide 25 mg tablets

SUMMARY:
The study was conducted as a open-label, balanced, randomized, two-treatment, two-period, two-sequence, single-dose, crossover, bioavailability study comparing Quinapril hydrochloride and Hydrochlorothiazide tablets 20 mg/25 mg of OHM Laboratories Inc (a subsidiary of Ranbaxy pharmaceuticals Inc) with AccureticTM tablets 20 mg/ 25 mg (containing quinapril hydrochloride 20 mg and hydrochlorothiazide 25 mg) manufactured by Parke Davis Pharmaceuticals Limited, Vega Baja, PR 00694, Made in Germany and distributed by Parke-Davis, Division of Pfizer Inc. NY, NY 10017 in healthy, adult, male, human subjects under fasting condition.

DETAILED DESCRIPTION:
Following an overnight fast of at least 10 hour, a single oral dose of Quinapril hydrochloride and Hydrochlorothiazide tablets 20 mg/25 mg or AccureticTM tablet 20 mg/ 25 mg (containing quinapril hydrochloride 20 mg and hydrochlorothiazide 25 mg) was administered during each period of the study, along with 240 mL of drinking water at ambient temperature and under low light condition and supervision of a trained study personnel.

A total of sixty-four (64) subjects were enrolled in the study. One subject (subject number 18) dropped out of the study and two subjects (subject number 47 and 50) were withdrawn from the study. Hence Sixty-one (61) subjects completed both the periods of the study.

For Quinapril and Hydrochlorothiazide pharmacokinetic and statistical analyses were performed on data from 61 subjects who completed both the periods of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Were in the age range of 18-45 years.
2. Were neither overweight nor underweight for their corresponding height as per the Life Insurance Corporation of India height/weight chart for non-medical cases.
3. Had voluntarily given written informed consent to participate in this study.
4. Were of normal health as determined by medical history and physical examination of the subjects performed within 21 days prior to the commencement of the study.

Exclusion Criteria:

1. History of allergy to quinapril, hydrochlorothiazide, sulfonamide derived drugs or related ACE inhibitors.
2. Subject who had sitting systolic blood pressure of less than 90 mmHg or >140 mmHg and diastolic blood pressure of less than 60 mmHg or > 90 mm Hg on the day of admission.
3. Any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations.
4. Presence of disease markers of HIV 1 or 2, Hepatitis B or C viruses or syphilis infection.
5. Presence of values which were significantly different from normal reference ranges and/or judged clinically significant for haemoglobin, total white blood cells count, differential WBC count or platelet count.
6. Positive for urinary screen testing of drugs of abuse (opiates or cannabinoids)
7. Presence of values which were significantly different from normal reference ranges and/or judged clinically significant for serum creatinine, blood urea nitrogen, serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT), serum alkaline phosphatase, serum bilirubin, plasma glucose or serum cholesterol.
8. Clinically abnormal chemical and microscopic examination of urine defined as presence of RBC, WBC (>4/HPF), epithelial cells (>4/HPF), glucose (positive) or protein (positive).
9. Clinically abnormal ECG or Chest X-ray.
10. History of serious gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological or haematological disease, diabetes or glaucoma.
11. History of any psychiatric illness which might impair the ability to provide written informed consent.
12. Regular smokers who smoked more than 10 cigarettes daily or had difficulty abstaining from smoking for the duration of each study period.
13. History of drug dependence or excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (1 unit equivalent to half pint of beer or 1 glass of wine or 1 measure of spirit) or had difficulty in abstaining for the duration of each study period.
14. Used any enzyme modifying drugs within 30 days prior to Day 1 of this study.
15. Participated in any clinical trial within 12 weeks preceding Day 1 of this study.
16. Subjects who, through completion of this study, had donated and/or lost more than 350 mL of blood in the past 3 months.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2007-10; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence evaluation of Ranbaxy Quinapril hydrochloride 20 mg and Hydrochlorothiazide 25 mg tablets under fasting conditions

CONTACTS AND LOCATIONS:
Locations (1):
- Ranbaxy Clinical Pharmacology Unit, Noida, Uttar Pradesh, India

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html